CLINICAL TRIAL: NCT03601091
Title: RANDOMİZED,DOUBLE-BLİND TRİAL OF EFFECT OF DEXMEDETOMİDİNE AND MİDAZOLAM SEDATİON ON HEART RATE VARİABİLİTY AFTER CORONARY ARTERY BYPASS GRAFT SURGERY
Brief Title: EFFECT OF DEXMEDETOMİDİNE AND MİDAZOLAM SEDATİON ON HEART RATE VARİABİLİTY AFTER CORONARY ARTERY BYPASS GRAFT SURGERY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, mustafa emre gürcü, Medical Doctor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/3/53
Record Dates: First submitted 2018-06-27; First posted 2018-07-26 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Effect of Sedation on Heart Rate Variability
Keywords: dexmedetomidine; coronary artery bypass graft; heart rate variability
MeSH Terms: interventions — Dexmedetomidine; Injections; Midazolam

STUDY DESIGN:
Intervention Model Description: RANDOMISED- DOUBLE BLINDED
Who Masked: Participant, Investigator
Masking Description: DOUBLE BLINDED
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PR (Active Comparator): PRECEDEX 200 mcg 2 ml,0,3 mcg/kg/h, intravenous continue infusion, 4 hours.
  Interventions: Drug: Precedex 200 MCG in 2 ML Injection
- DO (Active Comparator): DORMICUM 5MG/5 ML, 0,1 mg/kh/h, intravenous continue infusion for 4 hours
  Interventions: Drug: DORMICUM 5MG/5 ML

INTERVENTIONS:
Drug: Precedex 200 MCG in 2 ML Injection — Infusion therapy of the drug
  Arms: PR
Drug: DORMICUM 5MG/5 ML — Infusion therapy of the drug
  Arms: DO

SUMMARY:
The parasympathetic tone reduction and sympathetic tone enhancement, which are components of the autonomic nervous system (ANS) activity, increase the likelihood of malignant arrhythmias leading to ventricular fibrillation. Malignant arrhythmias are associated with high mortality and morbidity after coronary artery bypass graft (CABG) surgeries. Heart rate variability (HRV) is a physiological indicator of the effects of ANS activity on heart rate and is associated with a prognostic value for cardiac mortality. Dexmedetomidine has been shown to improve myocardial perfusion, reduce arrhythmia incidence, reduce inflammatory response, and reduce mortality in patients with coronary artery disease. The aim of this study investigate the effects of dexmedetomidine electrophysiologically on cardiac autonomic system by using HRV analysis for the purpose of sedation in patients who were followed up in the intensive care unit after coronary artery bypass graft surgery

DETAILED DESCRIPTION:
Malignant arrhythmias are associated with high mortality and morbidity after coronary artery bypass graft (CABG) operations. Heart rate variability (HRV) is a physiological indicator of the effects of activity on heart ANS rate and has prognostic value for cardiac mortality. Spectral analysis of HRV can provide an assessment of adrenergic and cholinergic system activities during anesthesia. With the "power spectral" analysis of HRV, important clinical information can be obtained about the effects of anesthesia on the autonomic nervous system and the central nervous system. Decrease in HRV has a prognostic value for cardiac-induced mortality. The disease, which is transferred to intensive care unit (ICU) after CABG, is sedated with different medicines until the time of extubation. One commonly used sedative drug is deksmedetomidine, an α2 receptor agonist. Alpha 2 (α2) receptor agonist drugs reduce myocardial oxygen consumption and heart rate with sympatholytic properties. Therefore, deksmedetomidine can be safely and effectively used in patients undergoing cardiac surgery without pro-tachyarrhythmic and / or negative inotropic effects.In this study, it was aimed to investigate electrophysiologic effects of cardiac autonomic system by using HRV analysis in dexmedetomine and midazolam patients who underwent elective CABG and were used for sedation in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre-operative normal sinus rhythm
* Ejection fraction (EF)> 45% on echocardiography (echocardiography) examination
* 25 and 65 years of age will be included.

Exclusion Criteria:

* Atrial fibrillation , atrial flutter, supraventricular tachycardia , AV block, ventricular extrasystole
* Cardiopulmonary bypass have been reported in patients with diabetes mellitus (DM),
* Chronic obstructive pulmonary disease (COPD),
* Previous cerebrovascular event will be excluded from the study.
* Patients receiving high-dose inotropic drug support after surgery (inotropic score of> 10 in the first 24 hours) and
* Patients re-operated for bleeding revision will be removed from the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 24 hours
  Low and high frequency of heart rate regarding with aritmia incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Emre Gurcu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided